CLINICAL TRIAL: NCT01243021
Title: Nurse Administered Early Warning Score System Can be Used for Emergency Department Triage
Brief Title: Validation of an Early Warning Score Based Triage System in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Dorthea Christensen, Bispebjerg Hospital, Anaestesiological Department
Other Study IDs: BBH98765
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
At Bispebjerg Hospital we have introduced an Early Warning Score based triage system , called Bispebjerg Early Warning Score (BEWS), in order to identify critically ill patient on arrival at the emergency department. The purpose of this study is to validate our triage system.

ELIGIBILITY:
Inclusion Criteria:

* "Red" patient
* Seen in our emergency department between 1. april 2009 and 30. september 2009

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: When arriving at the emergency department patients are divided into on of three groups (red, blue nd white) according to the severity of their condition based on common regional guidelines. Red patients are the most servelery ill or injured patients. A random sample of "red" patients are included in this study
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Critical illness | 48 hours
  The investigators have defined a critically ill patient as a patient who dies within 48 hours of arrival at the emergency department or who is admitted to ICU within 48 hours of arrival at the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Dorthea Christensen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

REFERENCES:
- [Derived] Christensen D, Jensen NM, Maaloe R, Rudolph SS, Belhage B, Perrild H. Nurse-administered early warning score system can be used for emergency department triage. Dan Med Bull. 2011 Jun;58(6):A4221. PMID 21651873